CLINICAL TRIAL: NCT05440162
Title: Prevelane and Short Term Outcome of Hypernatremic Dehydration in Children With Acute Gastroenteritis in Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aya Ahmed Mostafa, resident doctor at pediatric department at faculty of medicine sohag university hospital, Sohag University
Other Study IDs: Soh-Med-22-06-08
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Gastroenteritis Acute
MeSH Terms: interventions — Water-Electrolyte Balance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: electrolyte — follow up NA

SUMMARY:
Hypernatremic dehydration (HND) is a common and potentially life-threatening condition in children. It is defined by a serum level of sodium greater than or equal to 145 mmol/L . HND is a type of acute dehydration constitutes a medical emergency and requires a rapid diagnosis for adequate and quick management. It is characterized by a deficit of total body water (TBW) relative to total body sodium (TBS) levels due to either loss of free water, or excessive administration of hypertonic sodium solutions. It is common in infants. Net water loss as seen in diarrhea is the most common cause of hypernatremia. Clinical interventions at the hospital settings or accidental sodium loading usually cause hypertonic sodium gain. It is common in developing countries where gastroenteritis is a common problem.

Most children with hypernatremia are dehydrated and have the typical signs and symptoms as weight loss, decreased skin turgor, pale skin color, and dry mucous membranes. Hypernatremia, even without dehydration, cause central nervous system symptoms according to the degree of sodium elevation and the acuity of the increase. Patients are irritable, restless weak, and lethargic. Some infants have a high-pitched cry. Alert patients are very thirsty, although nausea and fever may be present.

HND can lead to neurological impairment due to brain shrinkage, which can tear cerebral blood vessels, leading to brain hemorrhage. Cerebral hemorrhages are the most serious complications of HND that can eventually lead to convulsions and even coma .

The first priority in managing a child with HND is to stop the ongoing water loss by treating the underlying cause. The next step is to restore the intravascular volume with isotonic fluid. Dehydration can be treated with oral, nasogastric, or intravenous fluids. The child is given a fluid bolus, usually 20 mL/kg of the isotonic solution, over about 20 to 30 minutes. More severe dehydration needs repeated boluses at a faster rate. After the fluid bolus is given, the signs of dehydration should be reassessed in order to confirm a complete rehydration. Fluid loss should not be corrected rapidly. Cerebral edema as well as convulsions is serious risks during rapid rehydration, so correction of deficit should be achieved slowly and gradually over 48 hours and should not be decreased to less than 12 mEq/L. To prevent cerebral edema and convulsion, individuals with hypernatremia should be managed in such a way that the reduction rate of serum sodium occurs at approximately 10 to 12 mmol/L/24 hr.

Cerebral edema and seizures can be consequences of rapid correction of serum sodium level in these patients in whom the rate of fluid and sodium administration are inappropriate

ELIGIBILITY:
Inclusion Criteria:

* Children with acute gastroenteritis who fulfill the following criteria:

  1. Age from one month up to 10 years.
  2. Large frequent stools.
  3. Symptoms and signs of dehydration.
  4. Serum sodium level ≧ 145 mmol/L.

Exclusion Criteria:

1. Parenteral diarrhea.
2. Gastroenteritis more than 14 days

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: will be taken from patients' parents or their caregivers including onset, course and duration of gastroenteritis; frequency, volume, consistency and contents of diarrhea; frequency, volume and contents of vomiting and manifestations of dehydration.
  Detailed clinical examination will be done with stress on signs of shock and dehydration including looking for thirsty, irritability, pinched look, sunken eyes, dry inner side of cheeks, abdominal distention, deep and rapid breathing, weak and thready pulse, falling blood pressure, reduced quantity of urine according to WHO dehydration assessment scale.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
sodium percentage | 1year

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mujawar NS, Jaiswal AN. Hypernatremia in the Neonate: Neonatal Hypernatremia and Hypernatremic Dehydration in Neonates Receiving Exclusive Breastfeeding. Indian J Crit Care Med. 2017 Jan;21(1):30-33. doi: 10.4103/0972-5229.198323. PMID 28197048
- [Background] Arampatzis S, Frauchiger B, Fiedler GM, Leichtle AB, Buhl D, Schwarz C, Funk GC, Zimmermann H, Exadaktylos AK, Lindner G. Characteristics, symptoms, and outcome of severe dysnatremias present on hospital admission. Am J Med. 2012 Nov;125(11):1125.e1-1125.e7. doi: 10.1016/j.amjmed.2012.04.041. Epub 2012 Aug 28. PMID 22939097
- [Background] Colletti JE, Brown KM, Sharieff GQ, Barata IA, Ishimine P; ACEP Pediatric Emergency Medicine Committee. The management of children with gastroenteritis and dehydration in the emergency department. J Emerg Med. 2010 Jun;38(5):686-98. doi: 10.1016/j.jemermed.2008.06.015. Epub 2009 Apr 5. PMID 19345549
- [Background] Robertson G, Carrihill M, Hatherill M, Waggie Z, Reynolds L, Argent A. Relationship between fluid management, changes in serum sodium and outcome in hypernatraemia associated with gastroenteritis. J Paediatr Child Health. 2007 Apr;43(4):291-6. doi: 10.1111/j.1440-1754.2007.01061.x. PMID 17444832